CLINICAL TRIAL: NCT02475785
Title: Evaluation of Mini Plates Anchorage in Conjunction With Forsus Fatigue Resistant Device for Correction of Skeletal Class II Malocclusion in Growing Subjects: A Randomized Controlled Trial
Brief Title: Evaluation of Mini Plates Anchorage With Forsus Fatigue Resistant Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sherif A. Elkordy (Other)
Responsible Party: Sponsor-Investigator, Sherif A. Elkordy, Dr, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU001
Record Dates: First submitted 2015-06-13; First posted 2015-06-19 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Malocclusion, Angle Class II, Division 1
Keywords: Forsus Fatigue Resistant Device; Class II; anchorage; FFRD; mini plates; fixed functional appliance
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- FFRD and mini plates group (Experimental): Upper will be bonded, levelled and aligned until reaching 0.019 x 0.025 ss archwires.
  2 Y shaped mini plates will be inserted in the mandibular symphysis Insertion of the FFRD with Direct application over the mandibular mini plates
  Interventions: Device: FFRD and mini plates group
- conventional FFRD (Active Comparator): Upper and lower arches will be bonded, levelled and aligned until reaching 0.019 x 0.025 ss archwires.
  Insertion of FFRD with application over the lower archwire
  Interventions: Device: Conventional FFRD
- untreated control group (No Intervention): Patients will be observed for an average duration of 6-8 months

INTERVENTIONS:
Device: FFRD and mini plates group — FFRD direct loading over mini plates inserted in the mandibular symphysis
  Other Names: Mini plates anchored FFRD
  Arms: FFRD and mini plates group
Device: Conventional FFRD — FFRD inserted between maxillary and mandibular arches with the pushrods placed distal to mandibular canines
  Other Names: Dental anchored FFRD
  Arms: conventional FFRD

SUMMARY:
The purpose of this study is to determine if the Forsus Fatigue resistant Device appliance with direct skeletal mini plates anchorage is capable of achievement of skeletal mandibular effects while preventing the excessive proclination of the lower incisors at the end of the treatment when compared to the conventional Forsus Fatigue resistant Device appliance applied to the upper and lower dental arches in female patients with skeletal Class II malocclusion

DETAILED DESCRIPTION:
1. Background:

   Class II malocclusions are characterized by an incorrect relationship between the maxillary and mandibular arches due to skeletal or dental problems or a combination of both. The prevalence of this malocclusion was recently found to be 20.6% in the Egyptian population in the age between 11 and 14 years with mandibular retrusion as its most common characteristic. It was also mentioned that other populations showed the predominance of the mandibular retrusion (80%) as opposed to only 20% expressing excessive maxillary development.

   Class II profiles attractiveness was previously investigated in the literature. It was found that patients, their peers, orthodontists and oral surgeons, rated subjects with Class I profiles as more attractive than others with Class II profiles. It was also reported that the profile of normal adolescent patients were more favorably perceived by laypersons than untreated Class II division 1 malocclusion subjects.

   In growing patients having Class II mandibular retrusion, functional orthopedic appliances are commonly used for mandibular advancement based on the concept of growth modification. However, two main problems appeared to compromise the desired treatment outcomes of these appliances; the need for patient cooperation and the lack of the possibility of combining their use with fixed appliance therapy in order to shorten treatment duration.

   Many systematic reviews and meta-analyses were recently performed in the literature answering the question of whether removable functional appliances (RFAs) produced skeletal effects for correction the skeletal discrepancy through inducing actual increase in mandibular dimensions. Most recently two systematic reviews concluded that the skeletal effects of RFAs were minimal and could be considered of negligible clinical importance. They mentioned that treatment of Class II malocclusion with RFAs was associated with a minimal stimulation of mandibular growth, a minimal restriction of maxillary growth and more significant dento-alveolar and soft tissue changes.

   Fixed functional appliances were first introduced by Emil Herbst in 1905. Many types of fixed functional appliances were developed since then; including Jasper jumper and Twin force Bite corrector . The Forsus Fatigue Resistant Device (FFRD) was introduced by Bill Vogt in 2006. It represented a semi-rigid fixed functional alternative that was intended to overcome breakage problems of flexible fixed functional appliances. However, it was proven that dental changes were more significant than skeletal changes in the final occlusal results. These changes included mesial movement of the mandibular molars and proclination of the mandibular incisors. These unwanted tooth movements appeared to compromise the actual skeletal correction and jeopardize the stability of the results.

   Several attempts were proposed to counteract the unwanted dento-alveolar side effects of fixed functional appliances. Use of lingual arches, increase the dimensions of the archwires, the introduction of negative torque in the archwires and the use of lower incisor brackets with lingual crown torque are some examples. Some studies used the mini implants in an attempt to limit the unwanted dental effects of fixed functional appliances. These studies proved that mini implants anchorage reduced the lower incisors proclination but they in turn increased the upper incisors retroclination and were not able to achieve significant skeletal mandibular effects.

   Titanium mini plates were introduced for the use for orthodontic anchorage in 1999 as a skeletal anchorage system for open bite correction. They were proven to be well accepted by patients and providers, safe and effective adjunct for complex orthodontic cases. Other uses of mini plates in orthodontics included maxillary and mandibular molars distalization and orthodontic anchorage where it was reported that they were able to provide absolute anchorage. Bone anchored maxillary protraction using mini plates was reported to be successful in producing significant forward maxillary growth in Class III growing subjects. Recently mini plates were used for the direct loading of FFRD for correction of skeletal Class II malocclusion. They reported actual skeletal changes through the increase in the mandibular length with minimal dento-alveolar side effects. However, these results are only preliminary and have to be taken with caution because the study did not include control group.
2. Research Hypothesis:

   The null hypothesis (H0) of this research is that use of direct mini plate anchorage in conjunction with FFRD will not be able to induce skeletal rather than dental effects for correction of the skeletal Class II malocclusion in comparison with conventional FFRD therapy or with untreated growing Class II control subjects.
3. Objectives:

   The primary objective of this study is to determine if mini plates use in conjunction with FFRD will induce supplemental growth of the mandible in Class II malocclusion subjects with mandibular retrognathism.

   Secondary objectives include

   To determine if mini plates use in conjunction with FFRD will be able to:
   * Reduce the dento-alveolar side effects produced by fixed functional appliances in treatment of skeletal Class II subjects
   * Correct the soft tissue convexity in Class II subjects
   * Correct molar and canines relationships
   * Develop a patients' well-accepted treatment modality for correction of skeletal Class II malocclusion.
4. Study design

   According to the norms of the CONSORT STATEMENT, this study will be clinical with intervention, in which the allocation of the subjects will be randomized (block randomization). This study will be parallel with blinding for the outcome assessors. The primary purpose of this study will be treatment.
5. Participants - Settings and locations where the data are collected

   The treatment will be performed in the outpatient clinics of Department of Orthodontics of Cairo State University. This public university predominantly serves low-income population living in Cairo, Egypt. Data will be collected from April 2015 through August 2016.
6. Interventions

Two groups will receive treatment. Group 1 will be treated with the FFRD and mini plates anchorage for 10 months or until the correction of the malocclusion . Group 2 will be treated with conventional FFRD for 10 months or until the correction of the malocclusion. A third untreated control group will be included with an observation period of 6-8 months.

7a. Sample size

Our sample size calculation is based on a study which compared the use of Herbst appliance with and without mini implants anchorage and reported a significant increase in the Herbst mini screw group over their control group. The mean change in the mandibular length in the treatment and control groups were 4.6±2.43 mm and 0.9±2.09 mm respectively. Thus the mean difference was 3.7 with the within group standard deviation set at 2.26.

Because three groups will be compared, Bonferroni adjustment was used as alpha level/number of comparisons = 0.05/3= 0.0167 to adjust for multiple comparisons.

Power and Sample size calculation (PS) software (department of biostatistics Vanderbilt University) was used for sample size calculation. A t test was performed with the power was set as 0.9, allocation ratio of 1:1:1 and the Type I error probability (alpha) associated with this test was set as 0.0167. Results of the test showed that "The Group sample sizes of 11, 11 and 11 achieve 90% power to reject the null hypothesis of equal means with a significance level (alpha) of 0.0167"

Therefore, 33 subjects will be needed, with 11 subjects in each group. To account for patient loss to follow up (attrition), a sample size of 48 patients will be selected and divided into three groups, sixteen each.

7b. Interim analysis and stopping guidelines

In the group with mini plates anchorage, in case of mobility in the mini-plates in any subject, the load will be removed for about two weeks. After that, the load will be restored. If the mobility persists, surgical exposure of the mini plate will be done and either insertion of longer mini screws ion the same mini plate or a change in the position of the mini plate will be done.

Any harms, adverse effects or unintended effects of the study intervention will be documented and reported. Post-surgical swelling and pain are anticipated and will be addressed by antibiotics and pain killers. Other unanticipated surgical harms have to be immediately managed and will be reported. Harms related to the orthodontic appliances will be managed by the principal investigator.

8. Randomization

8a. Sequence generation

The randomization of the recruited subjects will be done with a randomized list, using random.org website. This list is made by an individual not involved in the clinical trial (S.B.)

8b. Type

The type of randomization will be block randomization. The number of blocks and block sizes will be blinded to the investigators.

9. Allocation and concealment mechanism

* Each patient will be allocated a number from sequentially numbered opaque sealed envelopes after fulfillment of the inclusion criteria and signing the informed consent to be enrolled in the study.
* According to the number, the patients will be then allocated into one of the groups using a randomization table.

  10. Implementation

Before the beginning of the research, the allocation sequence will be generated by a person not involved in the study (Dr S.B.). The random list will be sealed from the principal investigator who will enroll participants. After the participant takes a sealed number, S.B. will be contacted to implement the allocation. All the study contributors will have no access to the random list. The envelopes will be closed with the type of treatment selected for storage of the information.

11. Blinding

Blinding will be carried out only for the data assessment because the researchers, participants and subjects can not be blinded. Therefore, a person who does not know the nature of the trial will analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal Angle Class II division 1 malocclusion with a deficient mandible. (SNB ≤ 76°)
* Horizontal or neutral growth pattern. (MMP ≤ 30°)
* Increased overjet (min 5 mm) with Class II canine relationship. (minimum of half unit)
* Mandibular arch crowding less than 3 mm.
* At the time of insertion of the FFRD, the patients had to be in the "Middle Phalanx of the Middle finger" stage G or H (MP3 G or MP3 H stage) according to Rajagopal.

Exclusion Criteria:

* Systemic Disease.
* Any signs or symptoms or previous history of temporomandibular disorders (TMD) as clicking, crepitus, pain, limitation or deviation.
* Extracted or missing upper permanent tooth/teeth (except for third molars).
* Facial Asymmetry.
* Para-functional habits.
* Severe proclination or crowding that requires extractions in the lower arch.

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
correction of the skeletal Class II profile | expected average of 10 months
  This outcome will be detected through measurement of the mean change in the effective mandibular length and position from baseline data that when increased will result in a decrease in profile convexity. This measurement will be done after FFRD removal and correction of the sagittal relationship.
  Cone-beam computed tomography (CBCT) images will be used for analysis of this outcome where changes in effective mandibular length (Co-Gn) will be measured in mm

SECONDARY OUTCOMES:
Dento-alveolar side effects | expected average of 10 months
  The dento-alveolar side effects of the appliance therapy are to be detected. CBCT images will be used for analysis of this outcome where changes in the inclination and positions of incisors will be measured in degrees and mm respectively.
Angle of soft tissue convexity | expected average of 10 months
  Changes in the soft tissue angle of convexity will be detected by CBCT (in degrees) that contribute to soft tissue profile correction
Position of lips and Chin | expected average of 10 months
  Will be detected by CBCT; the position of the upper and lower lips and chin will be measured in mm relative to a frontal plane

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Elkordy, Phd, Principal Investigator — Associate Lecturer of Orthodontics Cairo University; Amr Abouelezz, MSc, Study Chair — Professor of Orthodontics Cairo University; Mona Fayed, Phd, Study Director — Associate Professor of Orthodontics Cairo University; Mai Abou el Fotouh, Phd, Study Director — Lecturer of Orthodontics Cairo University
Locations (1):
- Orthodontic department, Faculty of Oral and Dental Medicine, Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Pancherz H. Treatment of class II malocclusions by jumping the bite with the Herbst appliance. A cephalometric investigation. Am J Orthod. 1979 Oct;76(4):423-42. doi: 10.1016/0002-9416(79)90227-6. PMID 291343
- [Background] Pancherz H, Hansen K. Occlusal changes during and after Herbst treatment: a cephalometric investigation. Eur J Orthod. 1986 Nov;8(4):215-28. doi: 10.1093/ejo/8.4.215. No abstract available. PMID 3466794
- [Background] Sugawara J, Daimaruya T, Umemori M, Nagasaka H, Takahashi I, Kawamura H, Mitani H. Distal movement of mandibular molars in adult patients with the skeletal anchorage system. Am J Orthod Dentofacial Orthop. 2004 Feb;125(2):130-8. doi: 10.1016/j.ajodo.2003.02.003. PMID 14765050
- [Background] Umemori M, Sugawara J, Mitani H, Nagasaka H, Kawamura H. Skeletal anchorage system for open-bite correction. Am J Orthod Dentofacial Orthop. 1999 Feb;115(2):166-74. doi: 10.1016/S0889-5406(99)70345-8. PMID 9971928
- [Background] Celikoglu M, Unal T, Bayram M, Candirli C. Treatment of a skeletal Class II malocclusion using fixed functional appliance with miniplate anchorage. Eur J Dent. 2014 Apr;8(2):276-280. doi: 10.4103/1305-7456.130637. PMID 24966783
- [Background] Unal T, Celikoglu M, Candirli C. Evaluation of the effects of skeletal anchoraged Forsus FRD using miniplates inserted on mandibular symphysis: A new approach for the treatment of Class II malocclusion. Angle Orthod. 2015 May;85(3):413-9. doi: 10.2319/051314-345.1. Epub 2014 Oct 3. PMID 25279724
- [Background] Elkordy SA, Abouelezz AM, Fayed MM, Attia KH, Ishaq RA, Mostafa YA. Three-dimensional effects of the mini-implant-anchored Forsus Fatigue Resistant Device: A randomized controlled trial. Angle Orthod. 2016 Mar;86(2):292-305. doi: 10.2319/012515-55.1. Epub 2015 May 19. PMID 25989213
- [Background] Aslan BI, Kucukkaraca E, Turkoz C, Dincer M. Treatment effects of the Forsus Fatigue Resistant Device used with miniscrew anchorage. Angle Orthod. 2014 Jan;84(1):76-87. doi: 10.2319/032613-240.1. Epub 2013 Jun 17. PMID 23772682
- [Background] Phillips C, Griffin T, Bennett E. Perception of facial attractiveness by patients, peers, and professionals. Int J Adult Orthodon Orthognath Surg. 1995;10(2):127-35. PMID 9081998
- [Background] Bishara SE, Jakobsen JR. Profile changes in patients treated with and without extractions: assessments by lay people. Am J Orthod Dentofacial Orthop. 1997 Dec;112(6):639-44. doi: 10.1016/s0889-5406(97)70229-4. PMID 9423696
- [Background] El-Mangoury NH, Mostafa YA. Epidemiologic panorama of dental occlusion. Angle Orthod. 1990 Fall;60(3):207-14. doi: 10.1043/0003-3219(1990)0602.0.CO;2. PMID 2202237
- [Background] Tulloch JF, Proffit WR, Phillips C. Outcomes in a 2-phase randomized clinical trial of early Class II treatment. Am J Orthod Dentofacial Orthop. 2004 Jun;125(6):657-67. doi: 10.1016/j.ajodo.2004.02.008. PMID 15179390
- [Background] Koretsi V, Zymperdikas VF, Papageorgiou SN, Papadopoulos MA. Treatment effects of removable functional appliances in patients with Class II malocclusion: a systematic review and meta-analysis. Eur J Orthod. 2015 Aug;37(4):418-34. doi: 10.1093/ejo/cju071. Epub 2014 Nov 13. PMID 25398303
- [Background] Vogt W. The Forsus Fatigue Resistant Device. J Clin Orthod. 2006 Jun;40(6):368-77; quiz 358. No abstract available. PMID 16804253
- [Background] Heinig N, Goz G. Clinical application and effects of the Forsus spring. A study of a new Herbst hybrid. J Orofac Orthop. 2001 Nov;62(6):436-50. doi: 10.1007/s00056-001-0053-6. English, German. PMID 11765707
- [Background] Luzi C, Luzi V, Melsen B. Mini-implants and the efficiency of Herbst treatment: a preliminary study. Prog Orthod. 2013 Jul 31;14:21. doi: 10.1186/2196-1042-14-21. PMID 24325903
- [Background] Luzi C, Luzi V. [Skeletal Class II treatment with the miniscrew-anchored Herbst]. Orthod Fr. 2013 Dec;84(4):307-18. doi: 10.1051/orthodfr/2013070. Epub 2013 Nov 27. French. PMID 24280546
- [Background] Cornelis MA, Scheffler NR, Nyssen-Behets C, De Clerck HJ, Tulloch JF. Patients' and orthodontists' perceptions of miniplates used for temporary skeletal anchorage: a prospective study. Am J Orthod Dentofacial Orthop. 2008 Jan;133(1):18-24. doi: 10.1016/j.ajodo.2006.09.049. PMID 18174066
- [Background] De Clerck H, Cevidanes L, Baccetti T. Dentofacial effects of bone-anchored maxillary protraction: a controlled study of consecutively treated Class III patients. Am J Orthod Dentofacial Orthop. 2010 Nov;138(5):577-81. doi: 10.1016/j.ajodo.2009.10.037. PMID 21055597
- [Background] Kim S, Herring S, Wang IC, Alcalde R, Mak V, Fu I, Huang G. A comparison of miniplates and teeth for orthodontic anchorage. Am J Orthod Dentofacial Orthop. 2008 Feb;133(2):189.e1-9. doi: 10.1016/j.ajodo.2007.07.016. PMID 18249283
- [Background] Rajagopal R, Kansal S. A comparison of modified MP3 stages and the cervical vertebrae as growth indicators. J Clin Orthod. 2002 Jul;36(7):398-406. No abstract available. PMID 12165981